CLINICAL TRIAL: NCT01510210
Title: Identification of a Risk Profile to Guide Atrial Fibrillation Therapy
Brief Title: Risk Profile for Patients With Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.C. Van Gelder (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Sponsor-Investigator, I.C. Van Gelder, MD. PhD, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Other Study IDs: NHS2010B233
Record Dates: First submitted 2011-12-28; First posted 2012-01-16 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Arrhythmia; Rhythm control
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma stored at -80 degrees Celcius. If informed consent was obtained, DNA extraction has been performed.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to assess the risk profile in patients with atrial fibrillation, which represents the degree of changes in the atrial tissue and which can help predict in which patients rhythm control will be successful. This risk profile will consist of a combination of underlying (heart) disease and risk factors, measurements obtained from echocardiograms, and circulating biomarkers. Ultimately this risk profile can be used to guide type of rhythm control therapy in individual patients with atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation is responsible for substantial morbidity and mortality.Identification of patients with atrial fibrillation that is difficult to treat may improve the outcome of rhythm control therapy. Left atrial size could be a useful tool to select patients that will benefit from rhythm control therapy.Beside echocardiographic parameters,atrial fibrillation has been also associated with circulating biomarkers in blood like collagen metabolism, inflammatory mediators,neurohumoral factors and proteins/proteomic profiles. Beside more accepted risk factors (myocardial ischemia, diabetes and pulmonary disease)other less well-known clinical factors (sleep apnea, alcohol or other intoxication abuse, excessive physical activity, esophageal problems and increased body mass index) may also predict the outcome of rhythm control.It likes also plausible that recurrent atrial fibrillation within one month after start of rhythm control are associated with a different risk profile than late atrial fibrillation recurrence.During this study we will try to identify patients with atrial fibrillation who are more or less likely to respond to rhythm control therapy.

ELIGIBILITY:
Inclusion Criteria:

* Short-lasting symptomatic paroxysmal or persistent AF;
* Rhythm control strategy is preferred;
* No contra-indication for oral anticoagulation;
* Age > 18 years;
* Written informed consent

Exclusion Criteria:

* Total history of heart failure and/ or of severe valvular disease > 3 years;
* Severe valvular disease;
* Acute coronary syndrome/ myocardial infarction/ percutaneous coronary intervention/ coronary artery bypass surgery within the past one month;
* Post-operative AF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with short-lasting symptomatic paroxysmal or persistent AF
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Success of rhythm control | 12 month
  (1) < 1 second AF on end-of-study ECG; (2) < 30 seconds AF on end-of-study 48-hour Holter recording; (3) no AF on end-of-study 2 weeks Vitaphone ECG-card recording.

SECONDARY OUTCOMES:
Time to recurrence of (a)symptomatic AF | 1+3+6+9+12 month
  by assessment Percentage AF-burden on 24-holter during follow up
Failure of rhythm control, i.e. permanent AF | 1+3+6+9+12 month
  failure of rhythm control medication or electric cardioversion.
Risk profiles associated with early versus late AF recurrence | 1month and 12 month
  These parameters include underlying (heart) disease and risk factors (including age, family history for AF, signs of ischemia, coronary risk factors, pulmonary disease, diabetes, obesity, sleep apnea, esophageal problems), lifestyle (including caffeine and alcohol intake, exercise), autonomic trigger patterns of AF (i.e. vagal or adrenergic induced AF, or combination
Progression of paroxysmal AF to persistent or permanent AF and of persistent AF to permanent AF | 1+3+6+9+12 month
  clinical commplaints and 3-lead Holter monitoring will be used for assessing the onset of AF episode
Changes in atrial and ventricular echocardiographic parameters | 1month and 12 month
  Echocardiographic measures of LA size (LA size parasternal long axis view, LA volume,LA ejection fraction measurement, electro-echocardiographic parameters (Tissue Doppler total atrial conduction time (during sinus rhythm), AF cycle length and velocity (during AF)), and parameters of diastolic dysfunction, including E (early mitral valve flow velocity), A (late mitral valve flow velocity), E/A ratio, deceleration time, E' (early tissue Doppler lengthening velocity), and E/E' ratio
Cardiovascular morbidity and mortality | 1month and 12month
  hospitalization for cardiovascular reasons, non-cardiovascular and cardiovascular death will be carefully monitored through-out the study.
Pulmonary vein ablation | 1month, 3month, 6month, 9 month, 12month
  hospital admission for pulmonary vein ablation will be monitoring during the study.
Pathophysiological mechanisms associated with AF and success of rhythm control | baseline-12 months
  To study pathophysiological mechanisms of AF, e.g. collagen mediated or inflammation mediated AF

CONTACTS AND LOCATIONS:
Overall Officials: Harry Crijns, MD PhD, Principal Investigator — Maastricht University Medical Center; Isabelle C Van Gelder, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De With RR, Artola Arita V, Nguyen BO, Linz D, Ten Cate H, Spronk H, Schotten U, Jan van Zonneveld A, Erkuner O, Bayon MA, Schmidt AS, Luermans JGLM, Crijns HJGM, Van Gelder IC, Rienstra M. Different circulating biomarkers in women and men with paroxysmal atrial fibrillation: results from the AF-RISK and RACE V studies. Europace. 2022 Feb 2;24(2):193-201. doi: 10.1093/europace/euab179. PMID 34329401
- [Derived] Nguyen BO, Meems LMG, van Faassen M, Crijns HJGM, van Gelder IC, Kuipers F, Rienstra M. Gut-microbe derived TMAO and its association with more progressed forms of AF: Results from the AF-RISK study. Int J Cardiol Heart Vasc. 2021 May 24;34:100798. doi: 10.1016/j.ijcha.2021.100798. eCollection 2021 Jun. PMID 34095450
- [Derived] De With RR, Marcos EG, Dudink EAMP, Spronk HM, Crijns HJGM, Rienstra M, Van Gelder IC. Atrial fibrillation progression risk factors and associated cardiovascular outcome in well-phenotyped patients: data from the AF-RISK study. Europace. 2020 Mar 1;22(3):352-360. doi: 10.1093/europace/euz339. PMID 31865391